CLINICAL TRIAL: NCT01715545
Title: Availability of Poor Quality Embryos in Frozen-thawed Embryo Transfer Cycles
Brief Title: Availability of Poor Quality Embryos
Acronym: Availability
Status: Completed | Type: Observational
Sponsor: The Second Affiliated Hospital of Kunming Medical University (Other)
Responsible Party: Principal Investigator, Yang Jie, The Second Affiliated Hospital of Kunming Medical University, The Second Affiliated Hospital of Kunming Medical University
Other Study IDs: 200601YJ
Record Dates: First submitted 2012-10-24; First posted 2012-10-29 (Estimated); Last update posted 2012-10-29 (Estimated); Status verified 2012-10

CONDITIONS: Infertility
Keywords: day-3 poor quality embryo; vitrification; clinical outcome
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- day-3 poor quality embryos
- developmental stage: day3 poor quality embryos day4 morular day-5/6 blastocyst

SUMMARY:
The purpose of this study is to explore a method to identify the viability of day-3 poor quality embryos

DETAILED DESCRIPTION:
Day-3 poor quality embryos are related to significant lower clinical pregnancy,so freezing numerous poor quality embryos are clinical impractical. To ensure the successful pregnancy and to enhance the availability of the poor quality embryos, day-3 poor quality embryos are further cultured to different developmental stage and then cryopreserved. The viability of these embryos are tested in frozen-thawed transfer.

ELIGIBILITY:
Inclusion Criteria:

* unfertile women

Exclusion Criteria:

* women older than 40 years

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: unfertile women
Sampling Method: Non-Probability Sample
Enrollment: 481 (Actual)
Dates: Start 2011-01; Primary Completion 2012-04 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
pregnancy rate | 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jie Yang, Principal Investigator — The Second Affiliated Hospital of Kunming Medical University
Locations (1):
- The Second Affiliated Hospital of Kunming Medical University, Kunming, Yunnan, China

REFERENCES:
- [Background] (1) Lu LI, Xiao-xi SUN, Jun-ling CHEN, et al. Analysis of Factors Influencing Pregnancy Rate in Frozen-thawed Embryo Transfer. Journal of Reproduction and Contraception (2004) 15 (4):239-244